CLINICAL TRIAL: NCT01488175
Title: Clinical and Stereoradiological Comparison of the Results After Primary TKA Inserted With or Without the Use of a Tourniquet
Brief Title: Clinical and Stereoradiological Comparison of the Results After Primary Cemented Total Knee Arthroplasty Inserted With or Without the Use of a Tourniquet
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding problems
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Morten Grove Thomsen, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2-2011-100
Record Dates: First submitted 2011-12-02; First posted 2011-12-08 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis of the Knee
Keywords: TKA; RSA; Tourniquet; Arthroplasty; Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tourniquets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with tourniquet (Active Comparator)
  Interventions: Procedure: tourniquet
- without tourniquet (Placebo Comparator)
  Interventions: Procedure: no tourniquet

INTERVENTIONS:
Procedure: tourniquet — a tourniquet around the thigh is used during insertion of the TKA to achieve a bloodless environment
  Arms: with tourniquet
Procedure: no tourniquet — a tourniquet around the thigh is not used during insertion of the TKA
  Arms: without tourniquet

SUMMARY:
The purpose of this study is to investigate if the use of a tourniquet during insertion of a cemented primary total knee arthroplasty will influence clinical and radiological (measured with RSA X-ray technique) outcome.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis og osteoarthritis of the knee
* patients must be 18 years or older
* patients must understand and speak danish
* must be able to give signed consent

Exclusion Criteria:

* severe medical illness
* documented osteoporosis
* rheumatoid arthritis
* prior surgery in the knee
* neuropathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
migration of the prosthesis in millimeters assessed vith RSA. | 2 years
  does the use of a tourniquet around the thigh during insertion of a primary TKA affect postoperative migration of the prosthesis?

SECONDARY OUTCOMES:
postoperative pain. | 2 years
  Does the use of a tourniquet affect postoperative pain, patient satisfaciton and knee range of motion
Patient satisfaction (VAS-scale) | 2 years
  Does the use of a tourniquet affect postoperative pain, patient satisfaciton and knee range of motion
Knee range of motion (degrees) | 2 years
  Does the use of a tourniquet affect postoperative pain, patient satisfaciton and knee range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, M.D, Ph.D, Study Chair — Dept. of Orthopedics, University Hospital of Hvidovre, Denmark.
Locations (1):
- Dept. of Orthopedics, University Hospital of Hvidovre, Denmark., Hvidovre, Denmark